CLINICAL TRIAL: NCT05741476
Title: A Phase 3, Double-blind, Placebo-controlled, Randomized Study to Assess the Efficacy and Safety of Epicutaneous Immunotherapy With DBV712 250 μg in 4-7-year-old Children With Peanut Allergy (VITESSE)
Brief Title: Safety and Efficacy Study of Viaskin Peanut in Peanut-allergic Children 4-7 Years of Age
Acronym: VITESSE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V712-306 (VITESSE); EU CTIS (Other: 2022-502110-85-00)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Allergy, Peanut
Keywords: Peanut Hypersensitivity; Epicutaneous Immunotherapy (EPIT); Epicutaneous; Immunotherapy; Viaskin; Nut and Peanut Hypersensitivity; Food Hypersensitivity; Peanut Allergy; Food Allergy; Nut and Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Nut and Peanut Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DBPC Treatment Period: DBV712 250 mcg (Experimental): Participants will apply DBV712 250 mcg, epicutaneous system (or patch), daily for a period of 12 months. At Month 12, a post-treatment peanut DBPCFC will be performed, with a starting dose of 3 mg peanut protein with escalation to the highest dose of 1,000 mg peanut protein according to the following schedule: 3, 10, 30, 100, 300, 600, and 1,000 mg (2,043 mg cumulative dose).
  Interventions: Drug: DBV712
- DBPC Treatment Period: Placebo (Placebo Comparator): Participants will apply DBV712 matching placebo epicutaneous system (or patch), daily for a period of 12 months. At Month 12, a post-treatment peanut DBPCFC will be performed, with a starting dose of 3 mg peanut protein with escalation to the highest dose of 1,000 mg peanut protein according to the following schedule: 3, 10, 30, 100, 300, 600, and 1,000 mg (2,043 mg cumulative dose).
  Interventions: Other: Placebo
- Open Label Extension Period: DBV712 250 mcg (Experimental): Participants will apply DBV712 250 mcg, epicutaneous system (or patch), daily for a period of 2 additional years if they were randomized DBV712 250 mcg or for 3 years if they were randomized placebo. After 12 months of open-label treatment with DBV712 250 mcg, (i.e., at the end of Month 24), participants will undergo a peanut DBPCFC according to the following schedule: 3, 10, 30, 100, 300, 600, 1000, and 2000 mg (4043 mg cumulative dose). Participants who were randomized to placebo will also undergo an additional peanut DBPCFC after 24 months of open-label treatment with DBV712 250 mcg, (i.e., at the end of Month 36).
  Interventions: Drug: DBV712

INTERVENTIONS:
Drug: DBV712 — DBV712 250 mcg epicutaneous system.
  Other Names: ViaskinTM Peanut
  Arms: DBPC Treatment Period: DBV712 250 mcg
Other: Placebo — DBV712 matching placebo epicutaneous system.
  Arms: DBPC Treatment Period: Placebo
Drug: DBV712 — DBV712 250 mcg epicutaneous system.
  Other Names: ViaskinTM Peanut
  Arms: Open Label Extension Period: DBV712 250 mcg

SUMMARY:
The primary purpose of this study is to assess the efficacy and safety of daily DBV712 250 micrograms (mcg) to induce desensitization to peanut in peanut-allergic children 4-7 years of age over a 12-month double-blind, placebo-controlled (DBPC) Treatment Period.

DETAILED DESCRIPTION:
This study is consisting of a 4-week Screening Period, 12-month DBPC Treatment Period and an open-label extension of either 24 or 36-months duration so that each participant may have the opportunity to receive DBV712 for a total duration of 36 months. Following 36 months of treatment with DBV712 250 mcg, sustained unresponsiveness (SU) will be evaluated by subsequent open food challenge(s) [FC(s)] at 2-, 4-, and 6-months off treatment.

Maximum participant participation will be either approximately 44 or 56 months, depending on the participant's randomized treatment assignment. During the 4-week Screening Period, participants are required to meet 2 sequential screening parameters to determine eligibility prior to randomization:

* Assessment of peanut skin prick test (SPT) and serum peanut immunoglobulin-E (IgE)
* Peanut double-blind placebo-controlled food challenge (DBPCFC) to confirm peanut allergy and establish an entry peanut eliciting dose (ED). Participants with a peanut protein ED less than or equal to (≤) 100 milligram (mg) will be eligible for randomization.

The starting dose of the eligibility peanut DBPCFC will be 1 mg peanut protein and will escalate up to a highest single dose of 100 mg peanut protein (cumulative 144 mg) via the following schedule: 1, 3, 10, 30, 100 mg. Participants who react, with an eliciting dose (ED) (with dose-limiting symptoms) at or below the dose of 100 mg peanut protein will be considered eligible.

Randomization of eligible participants will occur in a 2:1 ratio to DBV712 250 mcg (active treatment) or placebo, respectively.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 4 through 7 years at Visit 1 (screening).
* Physician-diagnosed peanut allergy or children with a well-documented medical history of IgE-mediated reactions after ingestion of peanut and currently following a strict peanut-free diet.
* Peanut-specific IgE of >0.7 kilo allergy unit per liter (kUA/L) and a positive peanut SPT with the largest wheal diameter of ≥6 millimeter (mm) at Visit 1.
* An ED of ≤100 mg peanut protein at screening DBPCFC.

Participants may enter the Open-label Extension Period if they meet all of the following inclusion criteria:

* Signed ICF by the participant's parent(s)/caregiver(s). This consent should be signed after completion of the procedures in the randomized, DBPC Treatment Period, and before any procedure in Open-label Extension Period begins.
* Participants who perform the peanut DBPCFC at the end of Month 12 and have ≥80% compliance with investigational medicinal product (IMP).
* Parent(s)/caregiver(s) and participants willing to comply with all study requirements during the participant's participation in the study.

Key Exclusion Criteria:

* Severe generalized dermatologic disease involving the application area (interscapular region)
* Uncontrolled persistent asthma.
* Past or current immunotherapy for peanut allergy, including oral immunotherapy (OIT).
* Current immunotherapy for any allergen (including food allergy, allergic rhinitis and/or insect allergy), or treatment with any monoclonal antibody or biologic immunomodulatory therapy within 6 months prior to Visit 1.

Participants may not enter the Open-label Extension Period if they meet any of the following exclusion criteria:

* Participants who develop a severe anaphylactic reaction during the DBPCFC at the end of Month 12 with the event requiring tracheal intubation or leading to a cardiac arrest and/or to coma. Participants with other reported cases of severe anaphylaxis will be considered eligible to participate in the Open-label Extension Period, at the judgement of the Investigator.
* Any clinically significant disease which in the judgment of the Investigator may preclude safe participation or strict compliance with the protocol procedures.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
DBPC Treatment Period: Percentage of Treatment Responders in the DBV712 250 mcg Group Compared to Placebo Group | At Month 12
  A participant is defined as a treatment responder if: The initial ED was ≤30 mg peanut protein and the ED is ≥ 300 mg peanut protein at the post-treatment DBPCFC at Month 12; OR the initial ED was > 30 mg peanut protein and the ED is ≥600 mg peanut protein at the post-treatment DBPCFC at Month 12. Percentage of treatment responders in the DBV712 250 mcg group compared to the placebo group after 12 months of treatment in the target population will be reported.

SECONDARY OUTCOMES:
DBPC Treatment Period: Cumulative Reactive Dose (CRD) of Peanut Protein | At Month 12
  The Peanut Protein CRD is defined as the sum of all peanut protein doses taken by the participant during the DBPCFC (including the ED and any partial dose given before the reaction).
DBPC Treatment Period: Eliciting Dose (ED) of Peanut Protein | At Month 12
DBPC Treatment Period: Percentage of Participants with an Eliciting Dose (ED) ≥600 mg and ≥1,000 mg Peanut Protein at Month 12 | At Month 12
DBPC Treatment Period: Number of Participants by Maximum Severity of Allergic Reaction During the Peanut Oral Food Challenge | Baseline up to Month 12
  The maximum severity of allergic reaction will be assessed according to Consortium of Food Allergy Research (CoFAR) Grading Scale Version 3.0. The scale is Grade 1 (Mild) through 5, the higher the grade, the more severe the allergic reaction.

OTHER OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Adverse Events of Special Interest (AESI) | Screening up to 56 months.
  An AE: any untoward medical occurrence in a participant administered a study drug which may or may not have a causal relationship with the study drug. TEAEs were defined as AEs that developed or worsened or became serious during on- treatment period. A serious TEAE: any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. AESI defined as: Local AESIs- severe local site reactions; systemic AESIs systemic allergic reactions, including those leading to epinephrine use, whatever the causal relationship to IP; AEs leading to epinephrine or inhaled or systemic corticosteroid use irrespective of the causal relationship to IP. TEAE's will include physical examination, vital signs, AEs leading to topical corticosteroid use, assessment of pain.
Number of Participants With Systemic Allergic Reactions | Screening up to 56 months.
  Number of participants with systemic allergic reactions will be reported.
Total Score for Scoring Atopic Dermatitis (SCORAD) | Screening up to 56 months.
  SCORAD index is a clinical tool for assessing the severity of atopic dermatitis. Extent and intensity of eczema as well as subjective signs insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).

CONTACTS AND LOCATIONS:
Locations (79):
- United States (45):
  - DBV Investigative Site, Birmingham, Alabama
  - DBV Investigative Site, Tucson, Arizona
  - DBV Investigative Site, Little Rock, Arkansas
  - DBV Investigative Site, Los Angeles, California
  - DBV Investigative site, Mission Viejo, California
  - DBV Investigative Site, San Diego, California
  - DBV Investigative Site, San Francisco, California
  - DBV Investigative Site, San Jose, California
  - DBV Investigative Site, Aurora, Colorado
  - DBV Investigative Site, Colorado Springs, Colorado
  - DBV Investigative Site, Washington D.C., District of Columbia
  - DBV Investigative Site, Hollywood, Florida
  - DBV Investigative Site, Miami, Florida
  - DBV Investigative Site, St. Petersburg, Florida
  - DBV Investigative Site, Tampa, Florida
  - DBV Investigative site, Atlanta, Georgia
  - DBV Investigative Site, Marietta, Georgia
  - DBV Investigative Site, Chicago, Illinois
  - DBV Investigative Site, Normal, Illinois
  - DBV Investigative Site, Indianapolis, Indiana
  - DBV Investigative Site, Louisville, Kentucky
  - DBV Investigative Site, Baltimore, Maryland
  - DBV Investigative Site, Chevy Chase, Maryland
  - DBV Investigative Site, Boston, Massachusetts
  - DBV Investigative Site, Taunton, Massachusetts
  - DBV Investigative Site, Ann Arbor, Michigan
  - DBV Investigative Site, Ypsilanti, Michigan
  - DBV Investigative Site, Maplewood, Minnesota
  - DBV Investigative Site, Kansas City, Missouri
  - DBV Investigative Site, Great Neck, New York
  - DBV Investigative Site, New York, New York
  - DBV Investigative Site, Rochester, New York
  - DBV Investigative Site, Chapel Hill, North Carolina
  - DBV Investigative Site, Cincinnati, Ohio
  - DBV Investigative Site, Cleveland, Ohio
  - DBV Investigative Site, Columbus, Ohio
  - DBV Investigative Site, Philadelphia, Pennsylvania
  - DBV Investigative Site, Pittsburgh, Pennsylvania
  - DBV Investigative Site, Memphis, Tennessee
  - DBV Investigative Site, Nashville, Tennessee
  - DBV Investigative Site, Austin, Texas
  - DBV Investigative Site, Dallas, Texas
  - DBV Investigative Site, Houston, Texas
  - DBV Investigative Site, Seattle, Washington
  - DBV Investigative Site, Milwaukee, Wisconsin
- Australia (6):
  - DBV Investigative Site, Adelaide
  - DBV Investigative Site, Nedlands
  - DBV Investigative Site, Parkville
  - DBV Investigative Site, Richmond
  - DBV Investigative Site, South Brisbane
  - DBV Investigative Site, Westmead
- Canada (9):
  - DBV Investigative Site, Vancouver, British Columbia
  - DBV Investigative Site, Winnipeg, Manitoba
  - DBV Investigative Site, Burlington, Ontario
  - DBV Investigative Site, North York, Ontario
  - DBV Investigative Site, Ottawa, Ontario
  - DBV Investigative Site, Toronto, Ontario
  - DBV Investigative Site, Montreal, Quebec
  - DBV Investigative Site, Québec, Quebec
  - DBV Investigative Site, Hamilton
- France (6):
  - DBV Investigative Site, Angers
  - DBV Investigative Site, Brest
  - DBV Investigative Site, Bron
  - DBV Investigative Site, Nice
  - DBV Investigative Site, Strasbourg
  - DBV Investigative Site, Vandœuvre-lès-Nancy
- Germany (3):
  - DBV Investigative Site, Düsseldorf
  - DBV Investigative Site, Frankfurt
  - DBV Investigative Site, Ulm
- Ireland (2):
  - DBV Investigative Site, Cork
  - DBV Investigative Site, Dublin
- Netherlands (2):
  - DBV Investigative Site, Rotterdam
  - DBV Investigative Site, Utrecht
- Spain (2):
  - DBV Investigative Site, Madrid
  - DBV Investigative Site, Málaga
- United Kingdom (4):
  - DBV Investigative Site, London
  - DBV Investigative Site, Manchester
  - DBV Investigative Site, Sheffield
  - DBV Investigative Site, Southampton